CLINICAL TRIAL: NCT02558582
Title: Effect of Exercise Training in Arterial and Chronic Thromboembolic Pulmonary Hypertension in Switzerland and Standardization With European Countries
Brief Title: Effect of Exercise Training in Patients With Pulmonary Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-ZH-Nr. 2015-0231
Record Dates: First submitted 2015-09-14; First posted 2015-09-24 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary arterial hypertension; Chronic thromboembolic pulmonary hypertension; Rehabilitation; Oxygen
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Respiratory Rate; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Immediate Rehabilitation (Experimental): The PH specific rehabilitation consists of: bicycle ergometer training, respiratory training, dumbbell-training and (mental) gait training.
  Interventions: Behavioral: respiratory and exercise therapy
- Immediate Rehabilitation with oxygen (Experimental): The PH specific rehabilitation consists of: bicycle ergometer training, respiratory training, dumbbell-training and (mental) gait training.
  Patients who are not already under long-term oxygen therapy (LTOT) due to daytime hypoxemia will additionally be randomized to receive standardized supplemental oxygen therapy (SSOT) during training and nights.
  Interventions: Behavioral: respiratory and exercise therapy with supplemental oxygen
- Delayed Rehabilitation (Experimental): Waiting group that participates in the rehabilitation program after 3 months. The PH specific rehabilitation consists of: bicycle ergometer training, respiratory training, dumbbell-training and (mental) gait training.
  Interventions: Behavioral: respiratory and exercise therapy
- Delayed Rehabilitation with oxygen (Experimental): Waiting group that participates in the rehabilitation program after 3 months. The PH specific rehabilitation consists of: bicycle ergometer training, respiratory training, dumbbell-training and (mental) gait training.
  Patients who are not already under long-term oxygen therapy (LTOT) due to daytime hypoxemia will additionally be randomized to receive standardized supplemental oxygen therapy (SSOT) during training and nights.
  Interventions: Behavioral: respiratory and exercise therapy with supplemental oxygen

INTERVENTIONS:
Behavioral: respiratory and exercise therapy — The PH specific rehabilitation consists of: bicycle ergometer training, respiratory training, dumbbell-training and (mental) gait training.
  Arms: Delayed Rehabilitation; Immediate Rehabilitation
Behavioral: respiratory and exercise therapy with supplemental oxygen — The PH specific rehabilitation consists of: bicycle ergometer training, respiratory training, dumbbell-training and (mental) gait training.
  Patients who are not already under long-term oxygen therapy (LTOT) due to daytime hypoxemia will additionally be randomized to receive standardized supplemental oxygen therapy (SSOT) during training and nights.
  Arms: Delayed Rehabilitation with oxygen; Immediate Rehabilitation with oxygen

SUMMARY:
Pulmonary Hypertension (PH) is a serious disease with a dismal prognosis when left untreated. Advances in medical therapy have improved survival according to recent registries and systematic reviews, but are associated with high healthcare costs.

Earlier studies in Heidelberg, Germany showed good evidence for the effect of exercise training on improving exercise performance, quality of life and pulmonary hemodynamics in patients with pulmonary hypertension.

The main objectives of the present project are:

1. to investigate the quality of the implementation of a standardized 3 week in-hospital exercise training program on markers of outcome and disease severity in PH-patients in Switzerland immediately after training and after 3 and 12 month.
2. to look whether training with hyperoxia vs. standard care might be more effective.

This is a multicentre, randomized parallel-group trial where the intervention rehabilitation is delayed in one group so that they can serve as standard care controls for the others.

In a nested single-centre randomized-controlled trial patent will additionally be randomized to receive either usual rehabilitation (UR) or rehabilitation with standardized supplemental oxygen therapy (SSOT) during nights and ergometer training.

Patients will receive a PH specific rehabilitation program during 3 weeks followed by an instructed home-based training program for 12 weeks. Patients who are not already under long-term oxygen therapy (LTOT) due to daytime hypoxemia will additionally be randomized to receive standardized supplemental oxygen therapy (SSOT) during training and nights upon written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* WHO functional class II-IV
* PH diagnosed by right heart catheter showing:
* Baseline mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg
* Baseline pulmonary vascular resistance (PVR) > 240 dyn x s x cm-5
* Baseline pulmonary capillary wedge pressure (PCWP) ≤ 15 mm Hg
* Patients receiving maximal PH therapy including intensified treatment with diuretics and who have been stable for 2 months before entering the study
* PH target therapy should not be expected to change during the entire 15-week study period
* Negative pregnancy test (β-HCG) at the start of the trial
* Able to understand and willing to sign the Informed Consent Form

Exclusion Criteria:

* PH due to significant left heart disease (Wedge ≥ 15mmHg) or lung disease (FEV1 ≤ 60% predicted)
* Pregnancy at study onset
* Walking disability
* Any change in disease-targeted therapy within the last 2 months
* Any subject who is scheduled to receive another investigational drug during the course of this study
* Any other relevant concomitant disease
* Systolic blood pressure < 85 mmHg
* History or suspicion of inability to cooperate adequately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
6 Minute walking test | Change from Baseline to 15 weeks
Constant cardiopulmonary exercise testing change in endurance time | Change from Baseline to 15 weeks

SECONDARY OUTCOMES:
Quality of Life (questionnaire) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Minnesota living with heart failure questionnaire, Camphor, short form 36 item
Sit-to-Stand (physiological parameter) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Number of Sit-to-Stand performed in 1 minute
Stair Ascent (physiological parameter) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Force, Power and Time needed to climb 5 steps
Cognitive function (questionnaire) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Trail Making Test A & B, Stroop 1-3, 5 point test
Hemodynamic (physiological parameter) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Pulmonary artery pressure, cardiac output
Functional class (scale) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
Lung function (physiological parameter) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Forced vital capacity and liters in 1 second, Total lung capacity, diffusion of carbon dioxide
Daily activity (energy expenditure, steps per day, sleep time and efficiency, lying down time, physical activity level, metabolic equivalent units) | Baseline, 3 weeks, 15 weeks, 6 and 12 months
  Actigraphy

OTHER OUTCOMES:
Hospitalisation days | Baseline, 3 weeks, 15 weeks, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich Somaini, PD Dr., Principal Investigator — UniversityHospital Zurich
Locations (1):
- UniversityHospital Zurich, Department of Pulmonology, Zurich, Switzerland